CLINICAL TRIAL: NCT05867693
Title: Palmitoylethanolamide and Polydatin in Pediatric Irritable Bowel Syndrome: a Randomized Controlled Trial
Brief Title: Palmitoylethanolamide and Polydatin in Pediatric Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Di Nardo, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/ST/235
Record Dates: First submitted 2023-04-21; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — polydatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS patients assigned to palmithoylethanolamide/polydatin treatment (Experimental): Eligible patients (patients with symptoms meeting Rome IV criteria for diagnosis of IBS) will be randomly assigned to either co-micronised form palmithoylethanolamide/polydatin 200 mg/20 mg
  Interventions: Dietary Supplement: palmithoylethanolamide/polydatin
- IBS patients assigned to placebo treatment (Placebo Comparator): Eligible patients (patients with symptoms meeting Rome IV criteria for diagnosis of IBS) will be randomly assigned to Placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: palmithoylethanolamide/polydatin — Palmitoyl-ethanolamide, a saturated fatty acid amide of palmitic acid commonly found in egg yolk and peanuts, is chemically related to anandamide but exhibit low affinity for cannabinoid receptors, and participate in the control of inflammation and nociception mainly via down-regulation of mast cell activity. In addition, palmitoylethanolamide is able to reduce human colonic permeability both in vitro and in vivo. Interestingly, palmithoylethanolamide may act as mast cell modulator as a possible agonist for cannabinoid 2-like receptors; and as agonist for PPAR-α, transient receptor potential vanilloid type 1 (TRPV1), and 'orphan' G protein-coupled receptor 55.
  For these reasons, palmithoylethanolamide has emerged as potential regulators of nociception. Polydatin, a resveratrol glucoside, is a common dietary component derived from grapes which may act synergistically with palmithoylethanolamide in reducing mast cell activation and local oxidative stress.
  Arms: IBS patients assigned to palmithoylethanolamide/polydatin treatment
Dietary Supplement: placebo — After the screening phase, eligible patients will be randomly assigned to equivalent placebo
  Arms: IBS patients assigned to placebo treatment

SUMMARY:
This will be a randomised, double-blind, placebo-controlled, parallel-arm trial, designed to study the efficacy and safety of co-micronised palmithoylethanolamide/polydatin in pediatric patients (> 10 years) with Irritable bowel syndrome (IBS)

DETAILED DESCRIPTION:
The study will include a 2-week screening period, and a 12-week placebo-controlled treatment period . After the screening phase, eligible patients will be randomly assigned to either co-micronised form palmithoylethanolamide/polydatin 200 mg/20 mg, or the equivalent placebo (without the active treatment, replaced by equal amount of microcrystalline cellulose), three times a day, in a 1:1 ratio, for 12 weeks. Study visits were conducted every 4 weeks during the treatment period. All the subjects will be blindly allocated by means of scratch cards to one of the two treatment groups according to a computer-generated randomisation list provided by our statistician. A validated program will be used by an independent statistician to generate a randomisation list with blocks, block size = 4, pre-allocated to centres. Patients and study investigators will be blinded to the randomisation codes. The codes will be kept confidential until the end of the study when the randomisation code will be broken after the database lock.

After the screening visit and at the end of treatment all subjects will undergo intestinal permeability test and fecal calprotectin assay. Calprotectin assay will be performed using a commercially available enzyme-linked immunosorbent assay test (Calprest Eurospital, Trieste, Italy). According to the manufacturer, calprotectin levels exceeding 100 mg/kg were considered positive. Intestinal permeability will be evaluated using a liquid chromatography/mass spectrometry method previously published .

All subjects will undergo a formal clinical assessment and will be further phenotyped using validated questionnaires. Number of bowel movements per day and/or week and bowel habit characteristics, will be assessed by the Bristol stool scale.

The protocol will be approved by an independent ethics committee and conducted according to the Declaration of Helsinki and the principles of good clinical practice. The trial will be registered in a public registry.

The primary outcome will be the change in the abdominal pain symptoms (frequency and severity) according to validated score from baseline to the end of the treatment period. Secondary outcome will be modifications of intestinal permeability and fecal caprotectine.

ELIGIBILITY:
Inclusion Criteria:

* positive diagnosis of all IBS subtypes,
* negative fecal calprotectine
* nagative anti-transglutaminasi antibodies

Exclusion Criteria:

* Current use of nonsteroidal anti-infl ammatory drugs, corticosteroids and mast cell stabilisers
* Use of topical or systemic antibiotics in the last month,
* Continuous use of stimulant laxatives,
* Major abdominal surgery, inflammatory bowel disease, infectious diarrhoea, allergic diseases and other organic or psychiatric disorders.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-10-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
Change in the abdominal pain symptoms | 12 weeks
  The primary outcome will be the change in the abdominal pain symptoms (frequency and severity) according to validated score from baseline to the end of the treatment period. Secondary outcome will be modifications of intestinal permeability and fecal caprotectine.
  The primary outcome will be the change in the abdominal pain symptoms (frequency and severity) according to validated score from baseline to the end of the treatment period.

SECONDARY OUTCOMES:
Change in intestinal permeability | 12 weeks
  Secondary outcome will be modifications of intestinal permeability.Intestinal permeability will be evaluated using a liquid chromatography/mass spectrometry method.
Change in fecal calprotectin | 12 weeks
  Outcame 3 will be modification of fecal calprotectin. Calprotectin levels exceeding 100 mg/kg were considered positive

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Di Nardo, Prof, Study Chair — Sapienza University of Rome, Faculty of Medicine and Psychology, Sant'Andrea University Hospital
Locations (1):
- Prof Giovanni Di Nardo, Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No